CLINICAL TRIAL: NCT04604795
Title: A Randomized, Placebo Controlled, Double Blind, Single and Repeat Dose Escalation Phase 1 Study to Evaluate Safety, Tolerability, and Pharmacokinetics of GSK3915393 in Healthy Participants and Open Label Assessment of Coadministration of GSK3915393 With Grapefruit Juice and Itraconazole on the Pharmacokinetics of GSK3915393
Brief Title: Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of GSK3915393 in Healthy Participants and to Evaluate the Interaction Between GSK3915393 and Grapefruit Juice and Itraconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 213585
Record Dates: First submitted 2020-10-06; First posted 2020-10-27 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2022-06

CONDITIONS: Celiac Disease; Coeliac Disease
Keywords: Celiac disease; Itraconazole; Grape fruit juice; GSK3915393; Healthy Participants; Pharmacokinetics; First time into human
MeSH Terms: conditions — Celiac Disease | interventions — Itraconazole; Water

STUDY DESIGN:
Intervention Model Description: This is a 3-part study. Parts A and C will have a 5 period crossover design Part B will be conducted as a parallel group dose escalation study.
Who Masked: Participant, Investigator
Masking Description: Parts A and B will be double blind and Part C will be open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Part A:GSK3915393 DLs 1,3,4,intravenous (IV) microdose and placebo (Sequence A) (Experimental): In Part A, participants will receive dose levels (DLs) 1, 3, 4, IV microdose of GSK3915393, and placebo in a pre-determined sequence (Sequence A). There will be a washout period of at least 7 days between each dose. Oral dose levels will be determined based on safety, tolerability and PK data.
  Interventions: Drug: GSK3915393 Capsules; Drug: GSK3915393 Solution for Infusion; Drug: Placebo capsules
- Part A:GSK3915393 DLs 1,2,4,IV microdose and placebo (Sequence B) (Experimental): In Part A, participants will receive dose levels 1, 2, 4, IV microdose of GSK3915393 and placebo in a pre-determined sequence (Sequence B).
  There will be a washout period of at least 7 days between each dose. Oral dose levels will be determined based on safety, tolerability and PK data.
  Interventions: Drug: GSK3915393 Capsules; Drug: GSK3915393 Solution for Infusion; Drug: Placebo capsules
- Part A:GSK3915393 DLs 1,2,3,IV microdose and placebo (Sequence C) (Experimental): In Part A, participants will receive dose levels 1, 2, 3, IV microdose of GSK3915393 and placebo in a pre-determined sequence (Sequence C).
  There will be a washout period of at least 7 days between each dose. Oral dose levels will be determined based on safety, tolerability and PK data.
  Interventions: Drug: GSK3915393 Capsules; Drug: GSK3915393 Solution for Infusion; Drug: Placebo capsules
- Part A:GSK3915393 DLs 2,3,4,IV microdose and placebo (Sequence D) (Experimental): In Part A, participants will receive dose levels 2, 3, 4, IV microdose of GSK3915393 and placebo in a pre-determined sequence (Sequence D).
  There will be a washout period of at least 7 days between each dose. Oral dose levels will be determined based on safety, tolerability and PK data.
  Interventions: Drug: GSK3915393 Capsules; Drug: GSK3915393 Solution for Infusion; Drug: Placebo capsules
- Part B: Cohort 1: Participants receiving GSK3915393 DL X (Experimental): Participants will receive GSK3915393 dose level X twice daily during Part B of the study. Dose levels will be determined based on safety, tolerability and PK data from Part A.
  Interventions: Drug: GSK3915393 Capsules
- Part B: Cohort 1: Participants receiving placebo (Placebo Comparator): Participants will receive placebo matching GSK3915393 dose level X during Part B of the study.
  Interventions: Drug: Placebo capsules
- Part B: Cohort 2: Participants receiving GSK3915393 DL Y (Experimental): Participants will receive GSK3915393 dose level Y twice daily during Part B of the study. Dose levels will be determined based on safety, tolerability and PK data from Part A and Part B.
  Interventions: Drug: GSK3915393 Capsules
- Part B: Cohort 2: Participants receiving placebo (Placebo Comparator): Participants will receive placebo matching GSK3915393 dose level Y twice daily during Part B of the study
  Interventions: Drug: Placebo capsules
- Part B: Cohort 3: Participants receiving GSK3915393 DL Z (Experimental): Participants will receive GSK3915393 dose level Z twice daily during Part B of the study. Dose levels will be determined based on safety, tolerability and PK data from Part A and Part B.
  Interventions: Drug: GSK3915393 Capsules
- Part B: Cohort 3: Participants receiving placebo (Placebo Comparator): Participants will receive placebo matching GSK3915393 dose level Z twice daily during Part B of the study.
  Interventions: Drug: Placebo capsules
- Part C: GSK3915393 IV/GSK3915393 IV+ITZ/GSK3915393+water/GSK3915393+GFJ/GSK3915393+ITZ (Sequence A) (Experimental): Participants will receive GSK3915393 IV microdose in period 1 followed by combination of GSK3915393 IV microdose and itraconazole (ITZ) in period 2. Participants will then receive oral GSK3915393 plus water in period 3, oral GSK3915393 plus grape fruit juice (GFJ) in period 4 and oral GSK3915393 plus ITZ in period 5.
  Interventions: Drug: GSK3915393 Capsules; Drug: GSK3915393 Solution for Infusion; Drug: Itraconazole; Other: Water; Other: Grape fruit juice
- Part C: GSK3915393 IV/GSK3915393 IV+ITZ/GSK3915393+GFJ/GSK3915393+water/GSK3915393+ITZ (Sequence B) (Experimental): Participants will receive GSK3915393 IV microdose in period 1 followed by combination of GSK3915393 IV microdose and ITZ in period 2. Participants will then receive oral GSK3915393 plus GFJ in period 3, oral GSK3915393 plus water in period 4 and oral GSK3915393 plus ITZ in period 5.
  Interventions: Drug: GSK3915393 Capsules; Drug: GSK3915393 Solution for Infusion; Drug: Itraconazole; Other: Water; Other: Grape fruit juice

INTERVENTIONS:
Drug: GSK3915393 Capsules — GSK3915393 capsules will be given orally.
  Arms: Part A:GSK3915393 DLs 1,2,3,IV microdose and placebo (Sequence C); Part A:GSK3915393 DLs 1,2,4,IV microdose and placebo (Sequence B); Part A:GSK3915393 DLs 1,3,4,intravenous (IV) microdose and placebo (Sequence A); Part A:GSK3915393 DLs 2,3,4,IV microdose and placebo (Sequence D); Part B: Cohort 1: Participants receiving GSK3915393 DL X; Part B: Cohort 2: Participants receiving GSK3915393 DL Y; Part B: Cohort 3: Participants receiving GSK3915393 DL Z; Part C: GSK3915393 IV/GSK3915393 IV+ITZ/GSK3915393+GFJ/GSK3915393+water/GSK3915393+ITZ (Sequence B); Part C: GSK3915393 IV/GSK3915393 IV+ITZ/GSK3915393+water/GSK3915393+GFJ/GSK3915393+ITZ (Sequence A)
Drug: GSK3915393 Solution for Infusion — GSK3915393 solution for infusion will be administered intravenously.
  Arms: Part A:GSK3915393 DLs 1,2,3,IV microdose and placebo (Sequence C); Part A:GSK3915393 DLs 1,2,4,IV microdose and placebo (Sequence B); Part A:GSK3915393 DLs 1,3,4,intravenous (IV) microdose and placebo (Sequence A); Part A:GSK3915393 DLs 2,3,4,IV microdose and placebo (Sequence D); Part C: GSK3915393 IV/GSK3915393 IV+ITZ/GSK3915393+GFJ/GSK3915393+water/GSK3915393+ITZ (Sequence B); Part C: GSK3915393 IV/GSK3915393 IV+ITZ/GSK3915393+water/GSK3915393+GFJ/GSK3915393+ITZ (Sequence A)
Drug: Placebo capsules — Placebo matching GSK3915393 capsules will be given orally.
  Arms: Part A:GSK3915393 DLs 1,2,3,IV microdose and placebo (Sequence C); Part A:GSK3915393 DLs 1,2,4,IV microdose and placebo (Sequence B); Part A:GSK3915393 DLs 1,3,4,intravenous (IV) microdose and placebo (Sequence A); Part A:GSK3915393 DLs 2,3,4,IV microdose and placebo (Sequence D); Part B: Cohort 1: Participants receiving placebo; Part B: Cohort 2: Participants receiving placebo; Part B: Cohort 3: Participants receiving placebo
Drug: Itraconazole — Participants will be administered with GSK3915393 along with ITZ orally
  Arms: Part C: GSK3915393 IV/GSK3915393 IV+ITZ/GSK3915393+GFJ/GSK3915393+water/GSK3915393+ITZ (Sequence B); Part C: GSK3915393 IV/GSK3915393 IV+ITZ/GSK3915393+water/GSK3915393+GFJ/GSK3915393+ITZ (Sequence A)
Other: Water — Participants will be administered with GSK3915393 along with water orally
  Arms: Part C: GSK3915393 IV/GSK3915393 IV+ITZ/GSK3915393+GFJ/GSK3915393+water/GSK3915393+ITZ (Sequence B); Part C: GSK3915393 IV/GSK3915393 IV+ITZ/GSK3915393+water/GSK3915393+GFJ/GSK3915393+ITZ (Sequence A)
Other: Grape fruit juice — Participants will be administered with GSK3915393 along with GFJ orally
  Arms: Part C: GSK3915393 IV/GSK3915393 IV+ITZ/GSK3915393+GFJ/GSK3915393+water/GSK3915393+ITZ (Sequence B); Part C: GSK3915393 IV/GSK3915393 IV+ITZ/GSK3915393+water/GSK3915393+GFJ/GSK3915393+ITZ (Sequence A)

SUMMARY:
This is a 3-part first time into human study (FTIH) study for GSK3915393. Parts A and B of the study will evaluate the safety, tolerability and pharmacokinetics (PK) of single ascending and repeat oral doses of GSK3915393 in healthy adult participants. Part C will evaluate the impact of co-administration of GSK3915393 with grapefruit juice and itraconazole on the PK of GSK3915393.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 50 years of age inclusive, at the time of signing the informed consent.
* Healthy participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Negative coronavirus disease of 2019 (COVID-19) test on admission.
* Body weight >=40 kilograms (kg) and body mass index (BMI) within the range 18.5-29.9 kilograms per square meter (kg/m^2) (inclusive).
* Male or females: No restrictions for male participants. A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies: Is a woman of non-childbearing potential (WONCBP) OR Is a woman of childbearing potential (WOCBP) and using an acceptable contraceptive method from 30 days prior to first dose until follow up visit. The investigator should evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated in relationship to the first dose of study intervention). A WOCBP must have a negative highly sensitive pregnancy test (serum) at screening and on admission to the clinical unit. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or current evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal (Irritable bowel syndrome [IBS], Gastroesophageal reflux disease [GERD], nausea, vomiting or dysphagia), endocrine, hematological, neurological, or psychiatric disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Current evidence of active infection.
* Participants with signs/symptoms suggestive of COVID-19 (i.e. fever, cough, etc) within the past 14 days prior to screening and admission to clinical unit.
* Participants with known COVID-19 positive contacts in the past 14 days prior to screening and admission to clinical unit.
* Any history of suicidal behavior within the past 6 months or any history of attempted suicide in a participant's lifetime.
* Alanine transaminase (ALT) >1.5 times upper limit of normal (ULN).
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of gastrointestinal (GI) surgery (with exception of appendectomy).
* Average QT interval corrected using Fridericia's formula (QTcF) >450 milliseconds (msec) at screening.
* Any clinically relevant abnormality on the screening medical assessment, laboratory examination, or electrocardiogram.
* History of QTc prolongation, symptomatic cardiac arrhythmias or cardiac arrest.
* For Part C only, history of liver toxicity resulting from drug administration.
* For Part C only, history of intolerance to itraconazole.
* History of sensitivity to any of the study medication, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline Medical Monitor, contraindicates their participation.
* Use of any immunosuppressive medications within 6 months prior to entry.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, probiotics, antacids, herbal and dietary supplements (including Saint [St] John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half- lives (whichever is longer) prior to the first dose of study medication for each dosing, unless in the opinion of the Investigator and GlaxoSmithKline Medical Monitor the medication will not interfere with the study procedures or compromise participant safety. (Paracetamol is acceptable at a dose of no more than 500 milligrams [mg] at a time and no more than 2 grams [g] per day).
* Participants who have received a COVID-19 vaccine within 7 days of admission (or readmission) to the clinical unit or who are demonstrating signs/symptoms attributed to a COVID-19 vaccination that occurred greater than 7 days earlier.
* Recent donation of blood or blood products such that participation in the study would result in loss of blood in excess of 500 milliliter (mL) within 56 days.
* The participant has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dosing day.
* Unwillingness or inability to follow the procedures outlined in the protocol or any other type of medical research within 30 days of randomization.
* Presence of hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study treatment.
* Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* Positive Hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before dosing, or a positive drug screen reflecting consumption of illicit drugs.
* Regular alcohol consumption within 6 months prior to screening: An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Urinary cotinine levels indicative of smoking or use of tobacco or nicotine-containing products (e.g. nicotine patches or vaporizing devices) at screening or on admission to the unit.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 3-part study in healthy participants. Part A was a crossover design, single-dose (SD), Part B was a parallel group, repeat oral dose and Part C was a drug:drug interaction study.
Pre-assignment Details: Total 65 participants were enrolled at one center in United Kingdom. The dose escalation committee concluded that doses higher than 160 milligram (mg) once daily (QD) (Part A Period 4 dose) should not be given. Placebo arms across similar dosing strategies in Part B were combined as pre-specified in reporting and analysis plan.
Groups:
- PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg: Participants in Part A received a single oral dose of Placebo on Day 1 in treatment Period 1; followed by a single oral dose of GSK3915393 60 milligrams (mg) on Day 1 in treatment Period 2; followed by a single dose of GSK3915393 100 micrograms (mcg) intravenous (IV) on Day 1 in treatment Period 3; further followed by a single oral dose of GSK3915393 160 mg on Day 1 in treatment Period 4. Participants were dosed in the fed state. There was a washout period of 20 days between periods 1 and 2, washout period between treatment 2 and 3 was of 12 days, washout period between treatment periods 3 and 4 was of 20 days. There was a follow-up period of 14 days.
- Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg: Participants in Part A received a single oral dose of GSK3915393 15 mg on Day 1 in treatment Period 1; followed by a single oral dose of placebo on Day 1 in treatment Period 2; followed by a single dose of GSK3915393 100 mcg IV on Day 1 in treatment Period 3; further followed by a single oral dose of GSK3915393 160mg on Day 1 in treatment Period 4. Participants were dose in the fed state. There was a washout period of 20 days between periods 1 and 2, washout period between treatment 2 and 3 was of 12 days, washout period between treatment periods 3 and 4 was of 20 days. There was a follow-up period of 14 days.
- Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo: Participants in Part A received a single oral dose of GSK3915393 15 mg on Day 1 in treatment Period 1; followed by a single oral dose of GSK3915393 60 mg on Day 1 in treatment Period 2; followed by a single dose of GSK3915393 100 mcg IV on Day 1 in treatment Period 3; further followed by a single oral dose of placebo on Day 1 in treatment Period 4. Participants were dosed in fed state. There was a washout period of 20 days between Periods 1 and 2, washout period between treatment 2 and 3 was of 12 days, washout period between treatment periods 3 and 4 was of 20 days. There was a follow-up period of 14 days.
- Part A: GSK3915393 15mg/60mg/100mcg IV/160mg: Participants in Part A received a single oral dose of GSK3915393 15 mg on Day 1 in treatment Period 1; followed by a single oral dose of GSK3915393 60 mg on Day 1 in treatment Period 2; followed by a single dose of GSK3915393 100 mcg IV on Day 1 in treatment Period 3; further followed by a single oral dose of GSK3915393 160 mg on Day 1 in treatment Period 4. Participants were dosed in fed state. There was a washout period of 20 days between Period 1 and 2, washout period between treatment 2 and 3 was of 12 days, washout period between treatment period 3 and 4 was of 20 days. There was follow-up period of 14 days.
- Part B: Placebo: Participants received placebo matching with GSK3915393 as repeat oral dose for 14 days (dosing frequency twice a day [BID] or QD, matched to the frequency of dosing in the concurrent active treatment arm). The impact of food effect on pharmacokinetic (PK) of GSK3915393 was investigated following Ante-Meridiem (AM) dose on three days in all cohort (Day 3=fasted, Day 5= high fat breakfast, Day 7=standard breakfast).
- Part B: GSK3915393 20 mg (BID): Participants received GSK3915393 20 mg BID as repeat oral dose for 14 days. The impact of food effect on PK of GSK3915393 was investigated following AM dose on three days in all cohort (Day 3=fasted, Day 5= high fat breakfast, Day 7=standard breakfast).
- Part B: GSK3915393 80 mg (BID): Participants received GSK3915393 80 mg BID as repeat oral dose for 14 days. The impact of food effect on PK of GSK3915393 was investigated following AM dose on three days in all cohort (Day 3=fasted, Day 5= high fat breakfast, Day 7=standard breakfast).
- Part B: GSK3915393 160 mg (QD): Participants received GSK3915393 160 mg QD as repeat oral dose for 14 days. The impact of food effect on PK of GSK3915393 was investigated following AM dose on three days in all cohort (Day 3=fasted, Day 5= high fat breakfast, Day 7=standard breakfast).
- PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ: Participants in Part C received a single dose of GSK3915393 100 mcg IV on Day 1 in treatment Period 1; followed by a single dose of GSK3915393 100mcg IV along with Itraconazole (ITZ) on Day 1 in treatment Period 2; followed by a single oral dose of GSK3915393 20 mg along with grapefruit juice (GFJ) on Day 1 in treatment Period 3; followed by a single oral dose of GSK3915393 20mg along with water (WTR) on Day 1 in treatment Period 4; further followed by a single oral dose of GSK3915393 20 mg along with ITZ in treatment Period 5. There was a washout period of 6 days between treatment Periods 1 and 2, washout period of 24 days between treatment periods 2 and 3, washout period of 10 days between treatment periods 3 and 4 and washout period of 13 days between treatment periods 4 and 5. There was a follow-up of 14 days.
- Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ: Participants in Part C received a single dose of GSK3915393 100 mcg IV on Day 1 in treatment Period 1; followed by a single dose of GSK3915393 100 mcg IV along with ITZ on Day 1 in treatment Period 2; followed by a single oral dose of GSK3915393 20 mg+ water on Day 1 in treatment Period 3; followed by a single oral dose of GSK3915393 20mg along with GFJ on Day 1 in treatment Period 4; further followed by a single oral dose of GSK3915393 20 mg along with ITZ in treatment Period 5. There was a washout period of 6 days between treatment Periods 1 and 2, washout period of 24 days between treatment periods 2 and 3, washout period of 10 days between treatment periods 3 and 4 and washout period of 13 days between treatment periods 4 and 5. There was a follow-up of 14 days.
Period: Part A: Period 1 (Day 1)
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ
Started | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Washout Period 1(Up to Day 20)
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ
Started | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Period 2 (Day 1)
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ
Started | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
New Participant Enrolled and Dosed | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Washout Period 2 (Up to Day 12)
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ
Started | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Period 3 (Day 1)
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ
Started | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Washout Period 3 (Up to Day 20)
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ
Started | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Period 4 (Day 1)
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ
Started | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B: Up to Day 14
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ
Started | 0 | 0 | 0 | 0 | 10 | 10 | 9 | 9 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 8 | 9 | 9 | 9 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Period: Part C: Period 1 (Day 1)
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C: Washout Period 1 (Up to Day 6)
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Part C: Period 2 (Day 1)
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C: Washout Period 2 (Up to Day 24)
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C: Period 3 (Day 1)
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
New Participant Enrolled and Dosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C: Washout Period 3 (Up to Day10)
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Part C: Period 4 (Day 1)
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C: Washout Period 4 (Up to Day 13)
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Part C: Period 5 (Day 1)
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PartA: Placebo/GSK3915393 60mg/100mcg IV/160mg | Part A: GSK3915393 15mg/Placebo/100mcg IV/160mg | Part A: GSK3915393 15mg/60mg/100mcg IV/Placebo | Part A: GSK3915393 15mg/60mg/100mcg IV/160mg | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | PartC:GSK3915393 100mcg IV/100mcgIV+ITZ/20mg+GFJ/20+WTR/20+ITZ | Part C:GSK3915393 100mg IV/100mcgIV+ITZ/20mg+WTR/20+GFJ/20+ITZ | Total
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 10 | 10 | 9 | 9 | 6 | 7 | 65
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Between 19 and 65 years | 4 | 3 | 3 | 3 | 10 | 10 | 9 | 9 | 6 | 7 | 64
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 0 | 1 | 1 | 1 | 0 | 3 | 2 | 2 | 15
  Male | 2 | 1 | 3 | 2 | 9 | 9 | 9 | 6 | 4 | 5 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN - SOUTH EAST ASIAN HERITAGE | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
  BLACK OR AFRICAN AMERICAN | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 2 | 8
  WHITE -WHITE/CAUCASIAN/EUROPEAN HERITAGE | 3 | 2 | 3 | 2 | 9 | 9 | 5 | 8 | 4 | 4 | 49
  MIXED RACE | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  ASIAN -CENTRAL/SOUTH ASIAN HERITAGE | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
  ASIAN -EAST ASIAN HERITAGE | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With All Non-serious Adverse Events (AEs) and Serious AEs (SAEs) Following Administration of Oral Dose
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. SAE is defined as any serious adverse event that, at any dose which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, other situations as per investigator's medical or scientific judgment.
Time Frame: Up to 70 days
Population: Safety Population comprised of all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Placebo: Participants received a single oral dose of matching placebo on Day 1 in treatment Periods 1, 2 or 4.
- Part A: GSK3915393 15 mg: Participants received a single oral dose of GSK3915393 15 mg on Day 1 in treatment Period 1.
- Part A: GSK3915393 60 mg: Participants received a single oral dose of GSK3915393 60 mg on Day 1 in treatment Period 2.
- Part A: GSK3915393 160 mg: Participants received a single oral dose of GSK3915393 160 mg on Day 1 in treatment Period 4.
Arm/Group | Part A: Placebo | Part A: GSK3915393 15 mg | Part A: GSK3915393 60 mg | Part A: GSK3915393 160 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  All non-serious AEs | 1 | 2 | 3 | 1
  SAEs | 0 | 0 | 0 | 0

2. Primary Outcome: Part A: Number of Participants With Treatment-related AEs Following Administration of Oral Dose
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Number of participants with treatment related AEs were presented.
Time Frame: Up to 70 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK3915393 15 mg | Part A: GSK3915393 60 mg | Part A: GSK3915393 160 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Part B: Number of Participants With All Non-serious AEs and SAEs
Description: as for outcome 1
Time Frame: Up to 28 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 10 | 10 | 9 | 9
Participants
  All non-serious AEs | 3 | 5 | 1 | 5
  SAEs | 0 | 0 | 0 | 0

4. Primary Outcome: Part B: Number of Participants With Treatment-related AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Number of participants with treatment related AEs are presented.
Time Frame: Up to 28 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 10 | 10 | 9 | 9
Participants | 1 | 0 | 0 | 0

5. Primary Outcome: Part A: Number of Participants With Worst Case Chemistry Results by Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline Following Administration of Oral Dose
Description: Blood samples were collected for analysis of chemistry parameters. PCI ranges were >=2*Upper limit of normal (ULN) units per liter (U/L)(Alanine Aminotransferase [ALT]), >=2*ULN (U/L) (Aspartate Aminotransferase ([AST]), >=2*ULN (Alkaline Phosphatase [ALP]) (U/L), >=1.5*ULN (micromoles per liter) (bilirubin), <2 or >2.75 millimoles/liter (L) (mmol/L)(calcium), <3 or >11 mmol/L (glucose), <3 or >5.5 mmol/L (potassium), <130 or >150 mmol/L (sodium),<50 or >85 grams/liter (protein). Participants were counted in worst case category that their value changes to (low, within [w/in] range or no change [NC], or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, are recorded in 'To within Range No Change' category. Participants were counted twice if participant had values that changed 'To Low' and 'To High', so percentages may not add to 100 percentage (%).
Time Frame: Up to 70 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK3915393 15 mg | Part A: GSK3915393 60 mg | Part A: GSK3915393 160 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  ALT: To Low | 0 | 0 | 0 | 0
  ALT: To w/in Range or No change | 9 | 9 | 9 | 9
  ALT: To High | 0 | 0 | 0 | 0
  AST: To Low | 0 | 0 | 0 | 0
  AST: To w/in Range or No change | 9 | 9 | 9 | 9
  AST: To High | 0 | 0 | 0 | 0
  ALP: To Low | 0 | 0 | 0 | 0
  ALP: To w/in Range or No change | 9 | 9 | 9 | 9
  ALP: To High | 0 | 0 | 0 | 0
  Bilirubin: To Low | 0 | 0 | 0 | 0
  Bilirubin: To w/in Range or No change | 9 | 9 | 9 | 8
  Bilirubin: To High | 0 | 0 | 0 | 1
  Calcium: To Low | 0 | 0 | 0 | 0
  Calcium: To w/in Range or No change | 9 | 9 | 9 | 9
  Calcium: To High | 0 | 0 | 0 | 0
  Glucose: To Low | 0 | 0 | 0 | 0
  Glucose: To w/in Range or No change | 9 | 9 | 9 | 9
  Glucose: To High | 0 | 0 | 0 | 0
  Potassium: To Low | 0 | 0 | 0 | 0
  Potassium: To w/in Range or No change | 9 | 9 | 9 | 9
  Potassium: To High | 0 | 0 | 0 | 0
  Protein: To Low | 0 | 0 | 0 | 0
  Protein: To w/in Range or No change | 9 | 9 | 9 | 9
  Protein: To High | 0 | 0 | 0 | 0
  Sodium: To Low | 0 | 0 | 0 | 0
  Sodium: To w/in Range or No change | 9 | 9 | 9 | 9
  Sodium: To High | 0 | 0 | 0 | 0

6. Primary Outcome: Part A: Number of Participants With Worst Case Chemistry Results-creatinine by PCI Criteria Post-Baseline Relative to Baseline Following Administration of Oral Dose
Description: Blood samples were collected for analysis of creatinine. Participants were counted under increase of PCI if they had change from Baseline > 44.2 micromoles per Liter for any post Baseline assessment. Participants who did not meet this PCI criteria are counted as within (w/in) range.
Time Frame: Up to 70 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK3915393 15 mg | Part A: GSK3915393 60 mg | Part A: GSK3915393 160 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  W/in Range | 9 | 9 | 9 | 9
  Increase of PCI | 0 | 0 | 0 | 0

7. Primary Outcome: Part A: Number of Participants With Worst Case Chemistry Results-urea by PCI Criteria Post-Baseline Relative to Baseline Following Administration of Oral Dose
Description: Blood samples were collected for analysis of chemistry parameters. PCI range for Urea: High >10.5 mmol/L. Participants were counted in worst case category that their value changes to (within [w/in] range or no change [NC], or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, are recorded in 'To within Range No Change' category.
Time Frame: Up to 70 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK3915393 15 mg | Part A: GSK3915393 60 mg | Part A: GSK3915393 160 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  To w/in Range or No change | 9 | 9 | 9 | 9
  To High | 0 | 0 | 0 | 0

8. Primary Outcome: Part A: Number of Participants With Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline Following Administration of Oral Dose
Description: Blood samples were collected for analysis of hematology parameters. PCI ranges were >1*10^9 cell per liter (cells/L) (eosinophils), <0.2 or >0.54 proportion of red blood cells in blood (hematocrit), <80 or >180 grams per liter(g/L) (hemoglobin), <3 or >20 x10^9 cells/L (leukocytes), <0.8*10^9 cells/L (lymphocytes), <1.5 or >16*10^9 cells/L (neutrophils) and <100 or >550*10^9 cells/L (platelets). Participants were counted in worst case category that their value changes to (low, within range or no change or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (for example [e.g.], High to High), or whose value became within range, were recorded in "To within Range or No Change" category. Participants were counted twice if participant has values that changed 'To Low' & 'To High', so the percentages may not add to 100%.
Time Frame: Up to 70 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK3915393 15 mg | Part A: GSK3915393 60 mg | Part A: GSK3915393 160 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Eosinophils: To Low | 0 | 0 | 0 | 0
  Eosinophils: To w/in Range or No change | 9 | 9 | 9 | 9
  Eosinophils: To High | 0 | 0 | 0 | 0
  Hematocrit: To Low | 0 | 0 | 0 | 0
  Hematocrit: To w/in Range or No change | 9 | 9 | 9 | 9
  Hematocrit: To High | 0 | 0 | 0 | 0
  Hemoglobin: To Low | 0 | 0 | 0 | 0
  Hemoglobin: To w/in Range or No change | 9 | 9 | 9 | 9
  Hemoglobin: To High | 0 | 0 | 0 | 0
  Leukocytes: To Low | 0 | 0 | 0 | 0
  Leukocytes: To w/in Range or No change | 9 | 9 | 9 | 9
  Leukocytes: To High | 0 | 0 | 0 | 0
  Lymphocytes: To Low | 0 | 0 | 0 | 0
  Lymphocytes: To w/in Range or No change | 9 | 9 | 9 | 9
  Lymphocytes: To High | 0 | 0 | 0 | 0
  Neutrophils: To Low | 0 | 0 | 0 | 1
  Neutrophils: To w/in Range or No change | 9 | 9 | 9 | 8
  Neutrophils: To High | 0 | 0 | 0 | 0
  Platelets: To Low | 0 | 0 | 0 | 0
  Platelets: To w/in Range or No change | 9 | 9 | 9 | 9
  Platelets: To High | 0 | 0 | 0 | 0

9. Primary Outcome: Part A: Number of Participants With Worst Case Vital Sign Results by PCI Criteria Post-Baseline Relative to Baseline Following Administration of Oral Dose
Description: Vital signs included diastolic blood pressure (DBP), systolic blood pressure (SBP), pulse rate (PR), body temperature, respiratory rate (RR) and were measured after resting for at least 5 minutes in semi-supine position. PCI ranges were, SBP (millimeters of mercury[mmHg]): <85 (low) or >160 (high), DBP (mmHg): <45 (low) or >100 (high), heart rate (beats per minute): <40 (low) or >110 (high), respiration rate (breaths per minute):<=8 (low) or >20 (high) and body temperature (degrees Celsius) <=35.5 (low) or >38.0 (high). Participants were counted in worst case category that their value changes to (low, within range or no change, or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, are recorded in 'To W/in Range No Change' category. Participants were counted twice if participant had values that changed 'To Low' and 'To High', so percentages may not add to 100%.
Time Frame: Up to 70 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK3915393 15 mg | Part A: GSK3915393 60 mg | Part A: GSK3915393 160 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  SBP: To Low | 0 | 0 | 0 | 0
  SBP: To w/in Range or No change | 9 | 9 | 9 | 9
  SBP: To High | 0 | 0 | 0 | 0
  DBP: To Low | 0 | 0 | 0 | 0
  DBP: To w/in Range or No change | 9 | 9 | 9 | 9
  DBP: To High | 0 | 0 | 0 | 0
  PR: To Low | 0 | 0 | 0 | 0
  PR: To w/in Range or No change | 9 | 9 | 9 | 9
  PR: To High | 0 | 0 | 0 | 0
  Body temperature: To Low | 0 | 0 | 0 | 0
  Body temperature: To w/in Range or No change | 9 | 9 | 9 | 9
  Body temperature: To High | 0 | 0 | 0 | 0
  RR: To Low | 0 | 0 | 0 | 0
  RR: To w/in Range or No change | 9 | 9 | 9 | 9
  RR: To High | 0 | 0 | 0 | 0

10. Primary Outcome: Part A: Number of Participants With Worst Case Post-Baseline Abnormal Electrocardiogram (ECG) Findings Following Administration of Oral Dose
Description: Twelve lead ECG was obtained using an ECG machine that automatically calculated the heart rate and measured QTc, PR, QRS intervals. Abnormal findings were categorized as clinically significant and not clinically significant. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for number of participants with worst case post-Baseline abnormal ECG findings have been presented.
Time Frame: Up to 70 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK3915393 15 mg | Part A: GSK3915393 60 mg | Part A: GSK3915393 160 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Abnormal: Not Clinically Significant | 2 | 3 | 1 | 0
  Clinically Significant | 0 | 0 | 0 | 0

11. Primary Outcome: Part A: Number of Participants With Abnormal Physical Examination Findings Following Administration of Oral Dose
Description: A full physical examination was performed which included, at a minimum, assessments of the Skin, Cardiovascular, Respiratory, Gastrointestinal and Neurological systems.
Time Frame: Up to 70 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK3915393 15 mg | Part A: GSK3915393 60 mg | Part A: GSK3915393 160 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 0 | 0 | 0 | 0

12. Primary Outcome: Part B: Number of Participants With Worst Case Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline Following Administration of Repeat Oral Dose of GSK3915393
Description: Blood samples were collected for analysis of chemistry parameters. PCI ranges were >=2*ULN (U/L)(ALT), >=2*ULN (U/L) (AST), >=2*ULN (ALP) (U/L), >=1.5*ULN (micromoles per liter) (bilirubin), <2 or >2.75 millimoles/liter (L) (mmol/L)(calcium), <3 or >11 mmol/L (glucose), <3 or >5.5 mmol/L (potassium), <130 or >150 mmol/L (sodium),<50 or >85 grams/liter (protein). Participants were counted in worst case category that their value changes to (low, within [w/in] range or no change [NC], or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, are recorded in 'To within Range No Change' category. Participants were counted twice if participant had values that changed 'To Low' and 'To High', so percentages may not add to 100 percentage (%).
Time Frame: Up to 28 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 10 | 10 | 9 | 9
Participants
  ALT: To Low | 0 | 0 | 0 | 0
  ALT: To w/in Range or No change | 10 | 10 | 9 | 9
  ALT: To High | 0 | 0 | 0 | 0
  AST: To Low | 0 | 0 | 0 | 0
  AST: To w/in Range or No change | 10 | 10 | 9 | 8
  AST: To High | 0 | 0 | 0 | 1
  ALP: To Low | 0 | 0 | 0 | 0
  ALP: To w/in Range or No change | 10 | 10 | 9 | 9
  ALP: To High | 0 | 0 | 0 | 0
  Bilirubin: To Low | 0 | 0 | 0 | 0
  Bilirubin: To w/in Range or No change | 10 | 10 | 9 | 9
  Bilirubin: To High | 0 | 0 | 0 | 0
  Calcium: To Low | 0 | 0 | 0 | 0
  Calcium: To w/in Range or No change | 10 | 10 | 9 | 9
  Calcium: To High | 0 | 0 | 0 | 0
  Glucose: To Low | 0 | 0 | 0 | 0
  Glucose: To w/in Range or No change | 10 | 10 | 9 | 9
  Glucose: To High | 0 | 0 | 0 | 0
  Potassium: To Low | 0 | 0 | 0 | 0
  Potassium: To w/in Range or No change | 10 | 10 | 9 | 9
  Potassium: To High | 0 | 0 | 0 | 0
  Protein: To Low | 0 | 0 | 0 | 0
  Protein: To w/in Range or No change | 10 | 10 | 9 | 9
  Protein: To High | 0 | 0 | 0 | 0
  Sodium: To Low | 0 | 0 | 0 | 0
  Sodium: To w/in Range or No change | 10 | 10 | 9 | 9
  Sodium: To High | 0 | 0 | 0 | 0

13. Primary Outcome: Part B: Number of Participants With Worst Case Chemistry Results-urea by PCI Criteria Post-Baseline Relative to Baseline Following Administration of Repeat Oral Dose of GSK3915393
Description: Blood samples were collected for analysis of chemistry parameters. PCI range for Urea: High >10.5 mmol/L. Participants were counted in worst case category that their value changes to (within [w/in] range or NC, or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, are recorded in 'To within Range No Change' category.
Time Frame: Up to 28 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 10 | 10 | 9 | 9
Participants
  To W/in Range or No Change | 10 | 10 | 9 | 9
  To High | 0 | 0 | 0 | 0

14. Primary Outcome: Part B: Number of Participants With Worst Case Chemistry Results-creatinine by PCI Criteria Post-Baseline Relative to Baseline Following Administration of Repeat Oral Dose
Description: Blood samples were collected for analysis of creatinine. Participants were counted under increase of PCI if they had change from Baseline > 44.2 micromoles per Liter for any post Baseline assessment. Participants who did not meet this PCI criteria are counted as w/in range. Participants whose laboratory value became within range, were recorded in 'To within Range' category.
Time Frame: Up to 28 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 10 | 10 | 9 | 9
Participants
  W/in Range | 10 | 10 | 9 | 9
  Increase of PCI | 0 | 0 | 0 | 0

15. Primary Outcome: Part B: Number of Participants With Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline Following Repeat Oral Dose of GSK3915393
Description: Blood samples were collected for analysis of hematology parameters. PCI ranges were 1*10^9 cell per liter (cells/L) (eosinophils), <0.2 or >0.54 proportion of red blood cells in blood (hematocrit), <80 or >180 grams per liter(g/L) (hemoglobin), <3 or >20 x10^9 cells/L (leukocytes), <0.8*10^9 cells/L (lymphocytes), <1.5 or >16*10^9 cells/L (neutrophils) and <100 or >550*10^9 cells/L (platelets). Participants were counted in worst case category that their value changes to (low, within range or no change or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (for example [e.g.], High to High), or whose value became within range, were recorded in "To within Range or No Change" category. Participants were counted twice if participant has values that changed 'To Low' & 'To High', so the percentages may not add to 100%.
Time Frame: Up to 28 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 10 | 10 | 9 | 9
Participants
  Eosinophils: To Low | 0 | 0 | 0 | 0
  Eosinophils: To w/in Range or No change | 10 | 10 | 9 | 9
  Eosinophils: To High | 0 | 0 | 0 | 0
  Hematocrit: To Low | 0 | 0 | 0 | 0
  Hematocrit: To w/in Range or No change | 10 | 10 | 9 | 9
  Hematocrit: To High | 0 | 0 | 0 | 0
  Hemoglobin: To Low | 0 | 0 | 0 | 0
  Hemoglobin: To w/in Range or No change | 10 | 10 | 9 | 9
  Hemoglobin: To High | 0 | 0 | 0 | 0
  Leukocytes: To Low | 0 | 0 | 1 | 0
  Leukocytes: To w/in Range or No change | 10 | 10 | 8 | 9
  Leukocytes: To High | 0 | 0 | 0 | 0
  Lymphocytes: To Low | 0 | 0 | 0 | 0
  Lymphocytes: To w/in Range or No change | 10 | 10 | 9 | 9
  Lymphocytes: To High | 0 | 0 | 0 | 0
  Neutrophils: To Low | 0 | 1 | 2 | 2
  Neutrophils: To w/in Range or No change | 10 | 9 | 7 | 7
  Neutrophils: To High | 0 | 0 | 0 | 0
  Platelets: To Low | 0 | 0 | 0 | 0
  Platelets: To w/in Range or No change | 10 | 10 | 9 | 9
  Platelets: To High | 0 | 0 | 0 | 0

16. Primary Outcome: Part B: Number of Participants With Worst Case Vital Sign Results by PCI Criteria Post-Baseline Relative to Baseline Following Repeat Oral Dose of GSK3915393
Description: Vital signs included DBP, SBP, PR, body temperature, RR and were measured after resting for at least 5 minutes in semi-supine position. PCI ranges were, SBP (mmHg): <85 (low) or >160 (high), DBP (mmHg): <45 (low) or >100 (high), heart rate (beats per minute): <40 (low) or >110 (high), respiration rate (breaths per minute):<=8 (low) or >20 (high) and body temperature (degrees Celsius) <=35.5 (low) or >38.0 (high). Participants were counted in worst case category that their value changes to (low, within range or no change, or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, are recorded in 'To W/in Range No Change' category. Participants were counted twice if participant had values that changed 'To Low' and 'To High', so percentages may not add to 100%.
Time Frame: Up to 28 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 10 | 10 | 9 | 9
Participants
  SBP: To Low | 0 | 0 | 0 | 0
  SBP: To w/in Range or No change | 10 | 10 | 9 | 9
  SBP: To High | 0 | 0 | 0 | 0
  DBP: To Low | 0 | 0 | 0 | 0
  DBP: To w/in Range or No change | 10 | 10 | 9 | 9
  DBP: To High | 0 | 0 | 0 | 0
  PR: To Low | 0 | 1 | 0 | 0
  PR: To w/in Range or No change | 9 | 9 | 9 | 9
  PR: To High | 1 | 0 | 0 | 0
  Body temperature: To Low | 0 | 1 | 0 | 0
  Body temperature: To w/in Range or No change | 10 | 9 | 9 | 9
  Body temperature: To High | 0 | 0 | 0 | 0
  RR: To Low | 0 | 0 | 0 | 0
  RR: To w/in Range or No change | 9 | 10 | 9 | 9
  RR: To High | 1 | 0 | 0 | 0

17. Primary Outcome: Part B: Number of Participants With Worst Case Post-Baseline Abnormal ECG Findings Following Repeat Oral Dose of GSK3915393
Description: as for outcome 10
Time Frame: Up to 28 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 10 | 10 | 9 | 9
Participants
  Abnormal: Not Clinically Significant | 3 | 5 | 0 | 1
  Clinically Significant | 1 | 0 | 1 | 0

18. Primary Outcome: Part B: Number of Participants With Abnormal Physical Examination Findings Following Administration of Repeat Oral Dose of GSK3915393
Description: as for outcome 11
Time Frame: Up to 28 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 10 | 10 | 9 | 9
Participants | 0 | 0 | 0 | 0

19. Primary Outcome: Part C: Maximum Observed Plasma Drug Concentration (Cmax) Following IV Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1 hour 5 minutes, 1 hour 10 minutes, 1 hours 20 minutes, 1 hour 40 minutes, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 10 hours post-dose
Population: Pharmacokinetic Population comprised of all participants in the safety population who had at least 1 non-missing pharmacokinetic assessment (Non-quantifiable [NQ] values were considered as non-missing values).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Part C: GSK3915393 100 mcg IV: Participants received GSK3915393 100 mcg as IV dose.
Arm/Group | Part C: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Nanogram per milliliter | 4.7220 (36.38)

20. Primary Outcome: Part C: Cmax of GSK3915393 Following IV Dose of GSK3915393+ITZ
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1 hour 5 minutes, 1 hour 10 minutes, 1 hours 20 minutes, 1 hour 40 minutes, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, and 60 hours post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Part C: GSK3915393 100 mcg IV+ITZ: Participants received GSK3915393 100 mcg as IV dose in combination with ITZ
Arm/Group | Part C: GSK3915393 100 mcg IV+ITZ
Number analyzed (Participants) | 11
Nanogram per milliliter | 7.8839 (23.80)

21. Primary Outcome: Part C: Cmax Following Oral Dose of GSK3915393 in Combination With Water, GFJ and ITZ
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393. For Part C: GSK3915393 20 mg+ Water and Part C: GSK3915393 20 mg+ GFJ, concentrations after 24 hours post-dose were expected to be non-quantifiable. Cmax was derived based on collected assessments (up to 24 hours for Part C: GSK3915393 20 mg+ Water and Part C: GSK3915393 20 mg+ GFJ, up to 60 hours for Part C: GSK3915393 20 mg+ ITZ). Only the quantifiable concentration time points were to be considered for assessment of pharmacokinetic parameters.
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 24, 36, 48 and 60 hours post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Part C: GSK3915393 20 mg+ Water: Participants received GSK3915393 20 mg as oral dose in combination with water.
- Part C: GSK3915393 20 mg+ GFJ: Participants received GSK3915393 20 mg as oral dose in combination with GFJ.
- Part C: GSK3915393 20 mg+ ITZ: Participants received GSK3915393 20 mg as oral dose in combination with ITZ
Arm/Group | Part C: GSK3915393 20 mg+ Water | Part C: GSK3915393 20 mg+ GFJ | Part C: GSK3915393 20 mg+ ITZ
Number analyzed (Participants) | 11 | 12 | 10
Nanogram per milliliter | 145.5638 (63.79) | 145.0510 (46.66) | 982.5433 (33.02)
Statistical Analysis 1: Comparison: Part C: GSK3915393 20 mg+ Water vs Part C: GSK3915393 20 mg+ GFJ; Test type: Other; Ratio of geometric mean = 1.05, 90% CI 2-sided [0.833 to 1.331] — Log transformed Cmax was analyzed using a mixed model with fixed effects for regimen and period, and participants as random effect
Statistical Analysis 2: Comparison: Part C: GSK3915393 20 mg+ Water vs Part C: GSK3915393 20 mg+ ITZ; Test type: Other; Ratio of geometric mean = 6.45, 90% CI 2-sided [4.916 to 8.474] — Log transformed Cmax was analyzed using a mixed model with regimen, period, and regimen by period as fixed effects and participants as random effect

22. Primary Outcome: Part C: Time to Maximum Observed Plasma Drug Concentration (Tmax) Following IV Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: as for outcome 19
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part C: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Hour | 0.98 [0.67 to 0.98]

23. Primary Outcome: Part C: Tmax of GSK3915393 Following IV Dose of GSK3915393+ITZ
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: as for outcome 20
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part C: GSK3915393 100 mcg IV+ITZ
Number analyzed (Participants) | 11
Hour | 0.98 [0.98 to 1.00]

24. Primary Outcome: Part C: Tmax of GSK3915393 Following Oral Dose of GSK3915393 in Combination With Water, GFJ and ITZ
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393. For Part C: GSK3915393 20 mg+ Water and Part C: GSK3915393 20 mg+ GFJ, concentrations after 24 hours post-dose were expected to be non-quantifiable. Tmax was derived based on collected assessments (up to 24 hours for Part C: GSK3915393 20 mg+ Water and Part C: GSK3915393 20 mg+ GFJ, up to 60 hours for Part C: GSK3915393 20 mg+ ITZ). Only the quantifiable concentration time points were to be considered for assessment of pharmacokinetic parameters.
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 24, 36, 48 and 60 hours post-dose
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part C: GSK3915393 20 mg+ Water | Part C: GSK3915393 20 mg+ GFJ | Part C: GSK3915393 20 mg+ ITZ
Number analyzed (Participants) | 11 | 12 | 10
Hour | 0.67 [0.33 to 1.50] | 1.50 [0.67 to 2.02] | 1.25 [0.67 to 2.00]

25. Primary Outcome: Part C: Area Under Curve up to the Last Measurable Concentration (AUCLST[0-10]) Following IV Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: as for outcome 19
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part C: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Nanogram*hour per milliliter | 5.0061 (41.94)

26. Primary Outcome: Part C: AUCLST(0-24) of GSK3915393 Following IV Dose of GSK3915393+ITZ
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1 hour 5 minutes, 1 hour 10 minutes, 1 hours 20 minutes, 1 hour 40 minutes, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, and 24 hours post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part C: GSK3915393 100 mcg IV+ITZ
Number analyzed (Participants) | 11
Nanogram*hour per milliliter | 13.3393 (32.67)

27. Primary Outcome: Part C: AUCLST(0-24) of GSK3915393 Following Oral Dose of GSK3915393 in Combination With Water, GFJ and ITZ
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 and 24 hours post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part C: GSK3915393 20 mg+ Water | Part C: GSK3915393 20 mg+ GFJ | Part C: GSK3915393 20 mg+ ITZ
Number analyzed (Participants) | 11 | 12 | 10
Nanogram*hour per milliliter | 153.8368 (60.22) | 223.1288 (52.85) | 2129.2407 (39.04)

28. Primary Outcome: Part C: AUC From Time Zero to Infinity (AUC[0-inf]) Following IV Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: as for outcome 19
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part C: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Nanogram*hour per milliliter | 5.0325 (41.95)

29. Primary Outcome: Part C: AUC(0-inf) of GSK3915393 Following IV Dose of GSK3915393+ITZ
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: as for outcome 20
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part C: GSK3915393 100 mcg IV+ITZ
Number analyzed (Participants) | 11
Nanogram*hour per milliliter | 13.4250 (32.63)

30. Primary Outcome: Part C: AUC(0-inf) of GSK3915393 Following Oral Dose of GSK3915393 in Combination With Water, GFJ and ITZ
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393. For Part C: GSK3915393 20 mg+ Water and Part C: GSK3915393 20 mg+ GFJ, concentrations after 24 hours post-dose were expected to be non-quantifiable. AUC(0-inf) was derived based on collected assessments (up to 24 hours for Part C: GSK3915393 20 mg+ Water and Part C: GSK3915393 20 mg+ GFJ, up to 60 hours for Part C: GSK3915393 20 mg+ ITZ). Only the quantifiable concentration time points were to be considered for assessment of pharmacokinetic parameters.
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 24, 36, 48 and 60 hours post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part C: GSK3915393 20 mg+ Water | Part C: GSK3915393 20 mg+ GFJ | Part C: GSK3915393 20 mg+ ITZ
Number analyzed (Participants) | 11 | 12 | 10
Nanogram*hour per milliliter | 155.5203 (59.89) | 225.0856 (52.73) | 2141.8345 (39.15)
Statistical Analysis 1: Comparison: Part C: GSK3915393 20 mg+ Water vs Part C: GSK3915393 20 mg+ GFJ; Test type: Other; Ratio of geometric mean = 1.53, 90% CI 2-sided [1.268 to 1.847] — AUC(0-inf) was analyzed using a mixed model with fixed effects for regimen and period, and participants as random effect
Statistical Analysis 2: Comparison: Part C: GSK3915393 20 mg+ Water vs Part C: GSK3915393 20 mg+ ITZ; Test type: Other; Ratio of geometric mean = 12.51, 90% CI 2-sided [10.141 to 15.423] — Log transformed AUC(0-inf) was analyzed using a mixed model with regimen, period, and regimen by period as fixed effects and participants as random effect

31. Primary Outcome: Part C: Apparent Terminal Half-life (t1/2) of GSK3915393 Following IV Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: as for outcome 19
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part C: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Hours | NA [NA to NA] — NA indicates that t1/2 cannot be calculated due to insufficient number of quantifiable pharmacokinetic (PK) values in the terminal phase

32. Primary Outcome: Part C: t1/2 of GSK3915393 Following IV Dose of GSK3915393+ITZ
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: as for outcome 20
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part C: GSK3915393 100 mcg IV+ITZ
Number analyzed (Participants) | 11
Hour | NA [NA to NA] — NA indicates that t1/2 cannot be calculated due to insufficient number of quantifiable PK values in the terminal phase

33. Primary Outcome: Part C: t1/2 of GSK3915393 Following Oral Dose of GSK3915393 in Combination With Water, GFJ and ITZ
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393. For Part C: GSK3915393 20 mg+ Water and Part C: GSK3915393 20 mg+ GFJ, concentrations after 24 hours post-dose were expected to be non-quantifiable. t1/2 was derived based on collected assessments (up to 24 hours for Part C: GSK3915393 20 mg+ Water and Part C: GSK3915393 20 mg+ GFJ, up to 60 hours for Part C: GSK3915393 20 mg+ ITZ). Only the quantifiable concentration time points were to be considered for assessment of pharmacokinetic parameters.
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 24, 36, 48 and 60 hours post-dose
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part C: GSK3915393 20 mg+ Water | Part C: GSK3915393 20 mg+ GFJ | Part C: GSK3915393 20 mg+ ITZ
Number analyzed (Participants) | 11 | 12 | 10
Hours | NA [NA to NA] — NA indicates that t1/2 cannot be calculated due to insufficient number of quantifiable PK values in the terminal phase | NA [NA to NA] — NA indicates that t1/2 cannot be calculated due to insufficient number of quantifiable PK values in the terminal phase | NA [NA to NA] — NA indicates that t1/2 cannot be calculated due to insufficient number of quantifiable PK values in the terminal phase

34. Secondary Outcome: Part A: Cmax Following Single Oral Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1.5, 2, 3, 4, 6, 10, 12, 14, 24 and 36 hours post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Part A: GSK3915393 15 mg: Participants received a single oral dose of GSK3915393 15 mg.
- Part A: GSK3915393 60 mg: Participants received a single oral dose of GSK3915393 60 mg.
- Part A: GSK3915393 160 mg: Participants received a single oral dose of GSK3915393 160 mg.
Arm/Group | Part A: GSK3915393 15 mg | Part A: GSK3915393 60 mg | Part A: GSK3915393 160 mg
Number analyzed (Participants) | 9 | 9 | 9
Nanogram per milliliter | 58.7910 (71.78) | 235.4331 (82.49) | 1246.2994 (54.12)

35. Secondary Outcome: Part A: Cmax Following Single IV Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1 hour 5 minutes, 1 hour 10 minutes, 1 hours 20 minutes, 1 hour 40 minutes, 2, 2.5, 3, 3.5, 4, 5 and 6 hours post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Part A: GSK3915393 100 mcg IV: Participants received single dose of GSK3915393 100 mcg IV.
Arm/Group | Part A: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Nanogram per milliliter | 4.3979 (35.65)

36. Secondary Outcome: Part A: Tmax Following Single Oral Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1.5, 2, 3, 4, 6, 10, 12, 14, 24 and 36 hours post-dose
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part A: GSK3915393 15 mg | Part A: GSK3915393 60 mg | Part A: GSK3915393 160 mg
Number analyzed (Participants) | 9 | 9 | 9
Hour | 1.50 [1.00 to 2.00] | 1.52 [0.68 to 3.00] | 1.50 [0.33 to 4.00]

37. Secondary Outcome: Part A: Tmax Following IV Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: as for outcome 35
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part A: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Hour | 0.98 [0.33 to 0.98]

38. Secondary Outcome: Part A: AUCLST(0-24) Following Single Oral Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1.5, 2, 3, 4, 6, 10, 12, 14, and 24 hours post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part A: GSK3915393 15 mg | Part A: GSK3915393 60 mg | Part A: GSK3915393 160 mg
Number analyzed (Participants) | 9 | 9 | 9
Nanogram*hour per milliliter | 113.7272 (103.13) | 424.6809 (52.89) | 2221.3816 (55.49)

39. Secondary Outcome: Part A: AUCLST(0-6) Following Single IV Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: as for outcome 35
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part A: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Nanogram*hour per milliliter | 4.4466 (31.95)

40. Secondary Outcome: Part A: AUC(0-inf) Following Single Oral Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1.5, 2, 3, 4, 6, 10, 12, 14, 24 and 36 hours post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part A: GSK3915393 15 mg | Part A: GSK3915393 60 mg | Part A: GSK3915393 160 mg
Number analyzed (Participants) | 9 | 9 | 9
Nanogram*hour per milliliter | 116.5279 (101.68) | 431.3298 (51.93) | 2235.3991 (55.18)

41. Secondary Outcome: Part A: AUC(0-inf) Following Single IV Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: as for outcome 35
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part A: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Nanogram*hour per milliliter | 4.4790 (32.03)

42. Secondary Outcome: Part A: t1/2 Following Single IV Dose of GSK3915393 100 mcg IV
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: as for outcome 35
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part A: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Hour | NA [NA to NA] — NA indicates that t1/2 cannot be calculated due to insufficient number of quantifiable PK values in the terminal phase

43. Secondary Outcome: Part A: Clearance (CL) Following Single IV Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: as for outcome 35
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part A: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Liters per hour | 22.7675 (31.56)

44. Secondary Outcome: Part A: Volume of Distribution (Vd) Following Single IV Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: as for outcome 35
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part A: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Liters | 30.7890 (27.51)

45. Secondary Outcome: Part A: Absolute Bioavailability (F) Following Single Oral Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393. Absolute bioavailability is the amount of drug from a formulation that reaches the systemic circulation relative to an IV dose. It was expressed as ratio was calculated as (AUC[0-inf] for oral divided by oral dose) divided by (AUC[0-inf] for IV/dose given as IV).
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1.5, 2, 3, 4, 6, 10, 12, 14, 24 and 36 hours post-dose
Population: Pharmacokinetic Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part A: GSK3915393 15 mg | Part A: GSK3915393 60 mg | Part A: GSK3915393 160 mg
Number analyzed (Participants) | 8 | 9 | 9
Ratio | 0.20 (69.6) | 0.18 (40.7) | 0.29 (38.4)

46. Secondary Outcome: Part A: Fraction of Drug Escaping Hepatic Metabolism (FH) Following Single Oral Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393. FH was expressed as ratio and was calculated as: 1 minus hepatic extraction ratio. Hepatic extraction ratio=hepatic blood clearance (milliliters per minute)/hepatic blood flow (milliliters per minute).
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1.5, 2, 3, 4, 6, 10, 12, 14, 24 and 36 hours post-dose
Population: Pharmacokinetic Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Ratio
Arm/Group | Part A: GSK3915393 15 mg | Part A: GSK3915393 60 mg | Part A: GSK3915393 160 mg
Number analyzed (Participants) | 8 | 9 | 9
Ratio | 0.5367 [0.435 to 0.699] | 0.4617 [0.384 to 0.690] | 0.5107 [0.384 to 0.699]

47. Secondary Outcome: Part A: Product of Fraction of Drug Absorbed and Fraction of Drug Escaping Gut Metabolism (FA*FG) Following Oral Dose of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393. Product of FA*FG was calculated as: (absolute bioavailability [F] divided by fraction of drug escaping hepatic metabolism [FH]).
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1.5, 2, 3, 4, 6, 10, 12, 14, 24 and 36 hours post-dose
Population: Pharmacokinetic Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Ratio
Arm/Group | Part A: GSK3915393 15 mg | Part A: GSK3915393 60 mg | Part A: GSK3915393 160 mg
Number analyzed (Participants) | 8 | 9 | 9
Ratio | 0.3062 [0.191 to 1.454] | 0.3814 [0.238 to 0.639] | 0.5563 [0.328 to 1.173]

48. Secondary Outcome: Part A: Number of Participants With All Non-serious AEs and SAEs Following Administration Administration of IV Dose of GSK3915393
Description: as for outcome 1
Time Frame: Up to 21 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Participants
  All non-serious AEs | 4
  SAEs | 0

49. Secondary Outcome: Part A: Number of Participants With Worst Case Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline Following Administration Administration of IV Dose of GSK3915393
Description: as for outcome 12
Time Frame: Up to 21 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Participants
  ALT: To Low | 0
  ALT: To w/in Range or No change | 12
  ALT: To High | 0
  AST: To Low | 0
  AST: To w/in Range or No change | 12
  AST: To High | 0
  ALP: To Low | 0
  ALP: To w/in Range or No change | 12
  ALP: To High | 0
  Bilirubin: To Low | 0
  Bilirubin: To w/in Range or No change | 12
  Bilirubin: To High | 0
  Calcium: To Low | 0
  Calcium: To w/in Range or No change | 12
  Calcium: To High | 0
  Glucose: To Low | 0
  Glucose: To w/in Range or No change | 12
  Glucose: To High | 0
  Potassium: To Low | 0
  Potassium: To w/in Range or No change | 12
  Potassium: To High | 0
  Protein: To Low | 0
  Protein: To w/in Range or No change | 12
  Protein: To High | 0
  Sodium: To Low | 0
  Sodium: To w/in Range or No change | 12
  Sodium: To High | 0

50. Secondary Outcome: Part A: Number of Participants With Worst Case Chemistry Results-creatinine by PCI Criteria Post-Baseline Relative to Baseline Following Administration Administration of IV Dose of GSK3915393
Description: Blood samples were collected for analysis of creatinine. Participants were counted under increase of PCI if they had change from Baseline >44.2 micromoles per Liter for any post Baseline assessment. Participants who did not meet this PCI criteria are counted as w/in range.
Time Frame: Up to 21 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Participants
  W/in Range | 12
  Increase of PCI | 0

51. Secondary Outcome: Part A: Number of Participants With Worst Case Chemistry Results-urea by PCI Criteria Post-Baseline Relative to Baseline Following Administration of IV Dose of GSK3915393
Description: as for outcome 7
Time Frame: Up to 21 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Participants
  To w/in Range or No change | 12
  To High | 0

52. Secondary Outcome: Part A: Number of Participants With Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline Following Administration of IV Dose of GSK3915393
Description: as for outcome 8
Time Frame: Up to 21 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Participants
  Eosinophils: To Low | 0
  Eosinophils: To w/in Range or No change | 12
  Eosinophils: To High | 0
  Hematocrit: To Low | 0
  Hematocrit: To w/in Range or No change | 12
  Hematocrit: To High | 0
  Hemoglobin: To Low | 0
  Hemoglobin: To w/in Range or No change | 12
  Hemoglobin: To High | 0
  Leukocytes: To Low | 0
  Leukocytes: To w/in Range or No change | 12
  Leukocytes: To High | 0
  Lymphocytes: To Low | 0
  Lymphocytes: To w/in Range or No change | 12
  Lymphocytes: To High | 0
  Neutrophils: To Low | 1
  Neutrophils: To w/in Range or No change | 11
  Neutrophils: To High | 0
  Platelets: To Low | 0
  Platelets: To w/in Range or No change | 12
  Platelets: To High | 0

53. Secondary Outcome: Part A: Number of Participants With Worst Case Vital Sign Results by PCI Criteria Post-Baseline Relative to Baseline Following IV Dose of GSK3915393
Description: as for outcome 16
Time Frame: Up to 21 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Participants
  SBP: To Low | 0
  SBP: To w/in Range or No change | 12
  SBP: To High | 0
  DBP: To Low | 0
  DBP: To w/in Range or No change | 12
  DBP: To High | 0
  PR: To Low | 0
  PR: To w/in Range or No change | 12
  PR: To High | 0
  Body temperature: To Low | 0
  Body temperature: To w/in Range or No change | 12
  Body temperature: To High | 0
  RR: To Low | 0
  RR: To w/in Range or No change | 12
  RR: To High | 0

54. Secondary Outcome: Part A: Number of Participants With Worst Case Post-Baseline Abnormal ECG Findings Following Administration of IV Dose of GSK3915393
Description: as for outcome 10
Time Frame: Up to 21 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Participants
  Abnormal: Not Clinically Significant | 7
  Clinically Significant | 0

55. Secondary Outcome: Part A: Number of Participants With Abnormal Physical Examination Findings Following Administration of IV Dose of GSK3915393
Description: as for outcome 11
Time Frame: Up to 21 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: GSK3915393 100 mcg IV
Number analyzed (Participants) | 12
Participants | 0

56. Secondary Outcome: Part B: Cmax(0-10) Following Dosing of GSK3915393 on Days 1 and 14
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Days 1 and 14: Pre-dose, 20, 40 minutes, 1, 1.5, 2, 3, 4, 6, and 10 hours post-dose
Population: Pharmacokinetic Population. Only those participants with data available at the indicated time points were analyzed (represented by n=X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Groups:
- Part B: GSK3915393 20 mg (BID): Participants received repeat oral dose of GSK3915393 20 mg BID.
- Part B: GSK3915393 80 mg (BID): Participants received repeat oral dose of GSK3915393 80 mg BID.
Arm/Group | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 10 | 9 | 9
Nanograms per milliliter
  Day 1, n=10, 9, 9 | 64.7843 (45.50) | 408.5572 (107.00) | 823.7704 (42.34)
  Day 14, n=9, 9, 9: number analyzed (Participants) | 9 | 9 | 9
  Day 14, n=9, 9, 9 | 95.4416 (93.47) | 820.5354 (67.59) | 1710.7385 (48.78)

57. Secondary Outcome: Part B: Cmax(10-24) Following Repeat Dose 20 mg and 80 mg of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Days 1 and 14: 10 hours, 10 hours 20 minutes, 10 hours 40 minutes, 12, 12.5 ,13, 14, 16, and 24 hours post-dose
Population: as for outcome 56
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID)
Number analyzed (Participants) | 10 | 9
Nanograms per milliliter
  Day 1, n=10, 9 | 32.2127 (48.16) | 338.2996 (85.59)
  Day 14, n=9, 9: number analyzed (Participants) | 9 | 9
  Day 14, n=9, 9 | 62.0235 (114.26) | 931.2098 (62.68)

58. Secondary Outcome: Part B: Cmax(10-24) Following Dose 160 mg (QD) of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Days 1 and 14: 10, 24 hours post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 9
Nanograms per milliliter
  Day 1 | NA (NA) — NA indicates data is not available as Cmax(10-24) could not be considered reliable because only a single PK time point was collected beyond 10 hours post-dose for 160 mg once daily on Day 1
  Day 14 | NA (NA) — NA indicates data is not available as Cmax(10-24) could not be considered reliable because only a single PK time point was collected beyond 10 hours post-dose for 160 mg once daily on Day 14

59. Secondary Outcome: Part B: Tmax(0-10) Following Dosing of GSK3915393 on Days 1 and 14
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Days 1 and 14: Pre-dose, 20, 40 minutes, 1, 1.5, 2, 3, 4, 6, and 10 hours post-dose
Population: as for outcome 56
Measure: Median (Full Range); unit: Hour
Arm/Group | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 10 | 9 | 9
Hour
  Day 1, n=10, 9, 9 | 1.2583 [1.000 to 3.017] | 1.0167 [0.667 to 3.000] | 1.5000 [0.667 to 3.017]
  Day 14, n=9, 9, 9: number analyzed (Participants) | 9 | 9 | 9
  Day 14, n=9, 9, 9 | 1.5000 [0.667 to 3.000] | 0.7500 [0.333 to 1.000] | 0.6833 [0.300 to 1.000]

60. Secondary Outcome: Part B: Tmax(10-24) Following Repeat Dose 20 mg BID and 80 mg BID of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Days 1 and 14: 10 hours, 10 hours 20 minutes, 10 hours 40 minutes, 12, 12.5 ,13, 14, 16, and 24 hours post-dose
Population: as for outcome 56
Measure: Median (Full Range); unit: Hour
Arm/Group | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID)
Number analyzed (Participants) | 10 | 9
Hour
  Day 1, n=10, 9 | 2.0000 [2.000 to 4.000] | 2.0000 [0.667 to 3.000]
  Day 14, n=9, 9: number analyzed (Participants) | 9 | 9
  Day 14, n=9, 9 | 2.0000 [0.667 to 6.133] | 0.6667 [0.350 to 0.700]

61. Secondary Outcome: Part B: Tmax(10-24) Following Dose 160 mg (QD) of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Days 1 and 14: 10, 24 hours post-dose
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 9
Hour
  Day 1 | NA [NA to NA] — NA indicates data is not available as Tmax(10-24) could not be considered reliable because only a single PK time point was collected beyond 10 hours post-dose for 160 mg once daily on Day 1
  Day 14 | NA [NA to NA] — NA indicates data is not available as Tmax(10-24) could not be considered reliable because only a single PK time point was collected beyond 10 hours post-dose for 160 mg once daily on Day 14

62. Secondary Outcome: Part B: AUCLST(0-10) Following Dosing of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Days 1 and 14: Pre-dose, 20, 40 minutes, 1, 1.5, 2, 3, 4, 6, and 10 hours post-dose
Population: as for outcome 56
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour per milliliter
Arm/Group | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 10 | 9 | 9
Nanograms*hour per milliliter
  Day 1, n=10, 9, 9 | 90.7283 (47.48) | 570.8621 (73.35) | 1268.9518 (34.85)
  Day 14, n=9, 9, 9: number analyzed (Participants) | 9 | 9 | 9
  Day 14, n=9, 9, 9 | 173.2096 (63.74) | 873.9352 (44.84) | 1670.9421 (36.52)

63. Secondary Outcome: Part B: AUCLST(0-24) Following Repeat Dose 20 mg BID and 80 mg BID of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Days 1 and 14: Pre-dose, 20 minutes, 40 minutes, 1, 1.5, 2, 3, 4, 6, 10, 10 hours 20 minutes, 10 hours 40 minutes, 12, 12.5 ,13, 14, 16, and 24 hours post-dose
Population: as for outcome 56
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour per milliliter
Arm/Group | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID)
Number analyzed (Participants) | 10 | 9
Nanograms*hour per milliliter
  Day 1, n=10, 9 | 193.1524 (48.59) | 1242.5500 (67.19)
  Day 14, n=9, 9: number analyzed (Participants) | 9 | 9
  Day 14, n=9, 9 | 342.1653 (62.25) | 1856.9207 (45.22)

64. Secondary Outcome: Part B: AUCLST(0-24) Following Dose of GSK3915393 160 mg (QD)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Days 1 and 14: Pre-dose, 20 minutes, 40 minutess, 1, 1.5, 2, 3 ,4, 6, 10 and 24 hours post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour per milliliter
Arm/Group | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 9
Nanograms*hour per milliliter
  Day 1 | 1314.7399 (34.62)
  Day 14 | 1738.3433 (36.02)

65. Secondary Outcome: Part B: AUC(10-24) Following Repeat Dose 20 mg BID and 80 mg BID of GSK3915393
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Days 1 and 14: 10 hours, 10 hours 20 minutes, 10 hours 40 minutes, 12, 12.5 ,13, 14, 16, and 24 hours post-dose
Population: as for outcome 56
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour per milliliter
Arm/Group | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID)
Number analyzed (Participants) | 8 | 9
Nanograms*hour per milliliter
  Day 1 | 115.2199 (52.85) | 666.5290 (62.91)
  Day 14 | 189.9773 (47.30) | 959.7659 (49.53)

66. Secondary Outcome: Part B: AUC(10-24) Following Repeat Dose of GSK3915393 160 mg (QD)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Days 1 and 14: 10 and 24 hours post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour per milliliter
Arm/Group | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 9
Nanograms*hour per milliliter
  Day 1 | NA (NA) — NA indicates data is not available as AUC(10-24) could not be considered reliable because only a single PK time point was collected beyond 10 hours post-dose for 160 mg once daily on Day 1
  Day 14 | NA (NA) — NA indicates data is not available as AUC(10-24) could not be considered reliable because only a single PK time point was collected beyond 10 hours post-dose for 160 mg once daily on Day 14

67. Secondary Outcome: Part B: Cmax(0-10) Following First Dosing of GSK3915393 on Days 3, 5 and 7 (for Food-effect Assessment)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Days 3, 5 and 7: Pre-dose, 20, 40 minutes, 1, 1.5, 2, 3, 4, 6 and 10 hours post-dose
Population: as for outcome 56
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour per milliliter
Arm/Group | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 10 | 9 | 9
Nanograms*hour per milliliter
  Day 3, n=10, 9, 9 | 125.5298 (76.57) | 819.8381 (99.60) | 1324.4415 (25.48)
  Day 5, n= 10, 9, 9 | 56.9187 (54.99) | 235.7608 (75.63) | 550.0071 (75.02)
  Day 7, n= 9, 9, 9: number analyzed (Participants) | 9 | 9 | 9
  Day 7, n= 9, 9, 9 | 77.0364 (48.64) | 355.0055 (104.08) | 805.5202 (28.13)
Statistical Analysis 1: Comparison: Part B: GSK3915393 20 mg (BID); Test type: Other; Ratio of geometric mean = 0.47, 90% CI 2-sided [0.318 to 0.693] — Day 5 (High fat meal) versus (vs) Day 3 (fasted)
Statistical Analysis 2: Comparison: Part B: GSK3915393 20 mg (BID); Test type: Other; Ratio of geometric mean = 0.60, 90% CI 2-sided [0.405 to 0.882] — Day 7 (Standard meal) vs Day 3 (fasted)
Statistical Analysis 3: Comparison: Part B: GSK3915393 80 mg (BID); Test type: Other; Ratio of geometric mean = 0.29, 90% CI 2-sided [0.194 to 0.427] — Day 5 (High fat meal) vs Day 3 (fasted)
Statistical Analysis 4: Comparison: Part B: GSK3915393 80 mg (BID); Test type: Other; Ratio of geometric mean = 0.43, 90% CI 2-sided [0.292 to 0.643] — Day 7 (Standard meal) vs Day 3 (fasted)
Statistical Analysis 5: Comparison: Part B: GSK3915393 160 mg (QD); Test type: Other; Ratio of geometric mean = 0.42, 90% CI 2-sided [0.280 to 0.617] — Day 5 (High fat meal) vs Day 3 (fasted)
Statistical Analysis 6: Comparison: Part B: GSK3915393 160 mg (QD); Test type: Other; Ratio of geometric mean = 0.61, 90% CI 2-sided [0.410 to 0.903] — Day 7 (Standard meal) vs Day 3 (fasted)

68. Secondary Outcome: Part B: Tmax(0-10) Following First Dosing of GSK3915393 on Days 3, 5 and 7 (for Food-effect Assessment)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Days 3, 5 and 7: Pre-dose, 20, 40 minutes, 1, 1.5, 2, 3, 4, 6 and 10 hours post-dose
Population: Pharmacokinetic Pharmacokinetic Population. Only those participants with data available at the indicated time points were analyzed (represented by n=X in category titles).
Measure: Median (Full Range); unit: Hour
Arm/Group | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 10 | 9 | 9
Hour
  Day 3, n=10, 9, 9 | 0.6667 [0.333 to 1.000] | 1.0000 [0.333 to 2.033] | 1.0000 [0.667 to 2.000]
  Day 5, n= 10, 9, 9 | 1.5000 [0.667 to 3.000] | 1.5167 [1.000 to 4.000] | 3.0000 [1.000 to 4.000]
  Day 7, n= 9, 9, 9: number analyzed (Participants) | 9 | 9 | 9
  Day 7, n= 9, 9, 9 | 1.5000 [0.667 to 3.000] | 1.5000 [1.000 to 3.000] | 1.5000 [0.717 to 2.000]

69. Secondary Outcome: Part B: AUCLST(0-10) Following First Dosing of GSK3915393 on Days 3, 5 and 7 (for Food-effect Assessment)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Days 3, 5 and 7: Pre-dose, 20, 40 minutes, 1, 1.5 ,2, 3, 4, 6 and 10 hours post-dose
Population: as for outcome 68
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 10 | 9 | 9
Nanogram*hour per milliliter
  Day 3, n=10, 9, 9 | 115.6796 (60.32) | 883.5828 (75.58) | 1571.0637 (25.05)
  Day 5, n= 10, 9, 9 | 120.0480 (56.72) | 698.9908 (61.80) | 1320.6847 (25.74)
  Day 7, n= 9, 9, 9: number analyzed (Participants) | 9 | 9 | 9
  Day 7, n= 9, 9, 9 | 135.3659 (49.21) | 754.3745 (69.11) | 1551.1980 (21.66)
Statistical Analysis 1: Comparison: Part B: GSK3915393 20 mg (BID); Test type: Other; Ratio of geometric mean = 1.02, 90% CI 2-sided [0.867 to 1.205] — Day 5 (High fat meal) vs Day 3 (fasted)
Statistical Analysis 2: Comparison: Part B: GSK3915393 20 mg (BID); Test type: Other; Ratio of geometric mean = 1.11, 90% CI 2-sided [0.941 to 1.308] — Day 7 (Standard meal) vs Day 3 (fasted)
Statistical Analysis 3: Comparison: Part B: GSK3915393 80 mg (BID); Test type: Other; Ratio of geometric mean = 0.79, 90% CI 2-sided [0.671 to 0.933] — Day 5 (High fat meal) vs Day 3 (fasted)
Statistical Analysis 4: Comparison: Part B: GSK3915393 80 mg (BID); Test type: Other; Ratio of geometric mean = 0.85, 90% CI 2-sided [0.724 to 1.007] — Day 7 (Standard meal) vs Day 3 (fasted)
Statistical Analysis 5: Comparison: Part B: GSK3915393 160 mg (QD); Test type: Other; Ratio of geometric mean = 0.84, 90% CI 2-sided [0.713 to 0.992] — Day 5 (High fat meal) vs Day 3 (fasted)
Statistical Analysis 6: Comparison: Part B: GSK3915393 160 mg (QD); Test type: Other; Ratio of geometric mean = 0.99, 90% CI 2-sided [0.837 to 1.165] — Day 7 (Standard meal) vs Day 3 (fasted)

70. Secondary Outcome: Part B: Trough Concentration (Ctau) Following Dose of 20 mg BID and 80 mg BID of GSK3915393 on Day 14
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Day 14: Pre-dose, 20, 40 minutes, 1, 1.5 ,2, 3, 4, 6, 10, 10 hour 20 minutes, 10 hours 40 minutes, 12, 12.5, 13, 14, 16 and 24 hours post-dose
Population: Pharmacokinetic Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID)
Number analyzed (Participants) | 9 | 9
Nanograms per milliliter | 1.8808 (1.35678) | 3.3181 (2.36137)

71. Secondary Outcome: Part B: Trough Concentration (Ctau) Following Dose of 160 mg of GSK3915393 on Day 14
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393.
Time Frame: Day 14: Pre-dose, 20, 40 minutes, 1, 1.5 ,2, 3, 4, 6, 10, and 24 hours post-dose
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Part B: GSK3915393 160 mg (QD)
Number analyzed (Participants) | 9
Nanograms per milliliter | 2.5423 (1.75889)

72. Secondary Outcome: Part C: Number of Participants With All Non-serious AEs and SAEs
Description: as for outcome 1
Time Frame: Up to 72 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- Part C: GSK3915393 100 mcg+ITZ: Participants received GSK3915393 100 mcg as oral dose in combination with ITZ
- Part C: GSK3915393 20mg+Water: Participants received GSK3915393 20 mg as oral dose in combination with water.
- Part C: GSK3915393 20mg+GFJ: Participants received GSK3915393 20 mg as oral dose in combination with GFJ.
- Part C: SK3915393 20 mg+ITZ: Participants received GSK3915393 20 mg as oral dose in combination with ITZ
Arm/Group | Part C: GSK3915393 100 mcg IV | Part C: GSK3915393 100 mcg+ITZ | Part C: GSK3915393 20mg+Water | Part C: GSK3915393 20mg+GFJ | Part C: SK3915393 20 mg+ITZ
Number analyzed (Participants) | 12 | 11 | 11 | 12 | 10
Participants
  All non-serious AEs | 5 | 2 | 3 | 2 | 2
  SAEs | 0 | 0 | 0 | 0 | 0

73. Secondary Outcome: Part C: Number of Participants With Treatment-related AEs Following Dose of GSK3915393
Description: as for outcome 4
Time Frame: Up to 72 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK3915393 100 mcg IV | Part C: GSK3915393 100 mcg+ITZ | Part C: GSK3915393 20mg+Water | Part C: GSK3915393 20mg+GFJ | Part C: SK3915393 20 mg+ITZ
Number analyzed (Participants) | 12 | 11 | 11 | 12 | 10
Participants | 3 | 2 | 1 | 0 | 0

74. Secondary Outcome: Part C: Number of Participants With Worst Case Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline Following Dose Administration of GSK3915393
Description: as for outcome 12
Time Frame: Up to 72 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK3915393 100 mcg IV | Part C: GSK3915393 100 mcg+ITZ | Part C: GSK3915393 20mg+Water | Part C: GSK3915393 20mg+GFJ | Part C: SK3915393 20 mg+ITZ
Number analyzed (Participants) | 12 | 11 | 11 | 12 | 10
Participants
  ALT: To Low | 0 | 0 | 0 | 0 | 0
  ALT: To w/in Range or No change | 12 | 11 | 11 | 12 | 10
  ALT: To High | 0 | 0 | 0 | 0 | 0
  AST: To Low | 0 | 0 | 0 | 0 | 0
  AST: To w/in Range or No change | 12 | 11 | 11 | 12 | 10
  AST: To High | 0 | 0 | 0 | 0 | 0
  ALP: To Low | 0 | 0 | 0 | 0 | 0
  ALP: To w/in Range or No change | 12 | 11 | 11 | 12 | 10
  ALP: To High | 0 | 0 | 0 | 0 | 0
  Bilirubin: To Low | 0 | 0 | 0 | 0 | 0
  Bilirubin: To w/in Range or No change | 12 | 11 | 11 | 12 | 10
  Bilirubin: To High | 0 | 0 | 0 | 0 | 0
  Calcium: To Low | 0 | 0 | 0 | 1 | 0
  Calcium: To w/in Range or No change | 12 | 11 | 11 | 11 | 10
  Calcium: To High | 0 | 0 | 0 | 0 | 0
  Glucose: To Low | 0 | 0 | 0 | 0 | 0
  Glucose: To w/in Range or No change | 12 | 11 | 11 | 12 | 10
  Glucose: To High | 0 | 0 | 0 | 0 | 0
  Potassium: To Low | 0 | 0 | 0 | 0 | 0
  Potassium: To w/in Range or No change | 12 | 11 | 11 | 12 | 10
  Potassium: To High | 0 | 0 | 0 | 0 | 0
  Protein: To Low | 0 | 0 | 0 | 0 | 0
  Protein: To w/in Range or No change | 12 | 11 | 11 | 12 | 10
  Protein: To High | 0 | 0 | 0 | 0 | 0
  Sodium: To Low | 0 | 0 | 0 | 0 | 0
  Sodium: To w/in Range or No change | 12 | 11 | 11 | 12 | 10
  Sodium: To High | 0 | 0 | 0 | 0 | 0

75. Secondary Outcome: Part C: Number of Participants With Worst Case Chemistry Results: Creatinine by PCI Criteria Post-Baseline Relative to Baseline Following Dose Administration of GSK3915393
Description: as for outcome 14
Time Frame: Up to 72 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK3915393 100 mcg IV | Part C: GSK3915393 100 mcg+ITZ | Part C: GSK3915393 20mg+Water | Part C: GSK3915393 20mg+GFJ | Part C: SK3915393 20 mg+ITZ
Number analyzed (Participants) | 12 | 11 | 11 | 12 | 10
Participants
  W/in Range | 12 | 11 | 11 | 12 | 10
  Increase of PCI | 0 | 0 | 0 | 0 | 0

76. Secondary Outcome: Part C: Number of Participants With Worst Case Chemistry Results: Urea by PCI Criteria Post-Baseline Relative to Baseline Following Dose Administration of GSK3915393
Description: Blood samples were collected for analysis of chemistry parameters. PCI range for Urea: High >10.5 mmol/L. Participants were counted in worst case category that their value changes to ( within [w/in] range or no change [NC], or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, are recorded in 'To within Range No Change' category.
Time Frame: Up to 72 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK3915393 100 mcg IV | Part C: GSK3915393 100 mcg+ITZ | Part C: GSK3915393 20mg+Water | Part C: GSK3915393 20mg+GFJ | Part C: SK3915393 20 mg+ITZ
Number analyzed (Participants) | 12 | 11 | 11 | 12 | 10
Participants
  To W/in Range or No Change | 12 | 11 | 11 | 12 | 10
  To High | 0 | 0 | 0 | 0 | 0

77. Secondary Outcome: Part C: Number of Participants With Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline Following Dose Administration of GSK3915393
Description: as for outcome 15
Time Frame: Up to 72 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK3915393 100 mcg IV | Part C: GSK3915393 100 mcg+ITZ | Part C: GSK3915393 20mg+Water | Part C: GSK3915393 20mg+GFJ | Part C: SK3915393 20 mg+ITZ
Number analyzed (Participants) | 12 | 11 | 11 | 12 | 10
Participants
  Eosinophils: To Low | 0 | 0 | 0 | 0 | 0
  Eosinophils: To w/in Range or No change | 12 | 11 | 11 | 12 | 10
  Eosinophils: To High | 0 | 0 | 0 | 0 | 0
  Hematocrit: To Low | 0 | 0 | 0 | 0 | 0
  Hematocrit: To w/in Range or No change | 12 | 11 | 11 | 12 | 10
  Hematocrit: To High | 0 | 0 | 0 | 0 | 0
  Hemoglobin: To Low | 0 | 0 | 0 | 0 | 0
  Hemoglobin: To w/in Range or No change | 12 | 11 | 11 | 12 | 10
  Hemoglobin: To High | 0 | 0 | 0 | 0 | 0
  Leukocytes: To Low | 0 | 0 | 0 | 0 | 0
  Leukocytes: To w/in Range or No change | 12 | 11 | 11 | 12 | 10
  Leukocytes: To High | 0 | 0 | 0 | 0 | 0
  Lymphocytes: To Low | 0 | 0 | 0 | 0 | 0
  Lymphocytes: To w/in Range or No change | 12 | 11 | 11 | 12 | 10
  Lymphocytes: To High | 0 | 0 | 0 | 0 | 0
  Neutrophils: To Low | 1 | 0 | 0 | 0 | 0
  Neutrophils: To w/in Range or No change | 11 | 11 | 11 | 12 | 10
  Neutrophils: To High | 0 | 0 | 0 | 0 | 0
  Platelets: To Low | 0 | 0 | 0 | 0 | 0
  Platelets: To w/in Range or No change | 12 | 11 | 11 | 12 | 10
  Platelets: To High | 0 | 0 | 0 | 0 | 0

78. Secondary Outcome: Part C: Number of Participants With Worst Case Vital Sign Results by PCI Criteria Post-Baseline Relative to Baseline Following Dose Administration of GSK3915393
Description: as for outcome 16
Time Frame: Up to 72 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK3915393 100 mcg IV | Part C: GSK3915393 100 mcg+ITZ | Part C: GSK3915393 20mg+Water | Part C: GSK3915393 20mg+GFJ | Part C: SK3915393 20 mg+ITZ
Number analyzed (Participants) | 12 | 11 | 11 | 12 | 10
Participants
  SBP: To Low | 0 | 0 | 0 | 0 | 0
  SBP: To w/in Range or No change | 12 | 11 | 11 | 12 | 10
  SBP: To High | 0 | 0 | 0 | 0 | 0
  DBP: To Low | 0 | 0 | 0 | 0 | 0
  DBP: To w/in Range or No change | 12 | 11 | 11 | 12 | 10
  DBP: To High | 0 | 0 | 0 | 0 | 0
  PR: To Low | 0 | 0 | 0 | 0 | 0
  PR: To w/in Range or No change | 11 | 11 | 11 | 12 | 10
  PR: To High | 1 | 0 | 0 | 0 | 0
  Temperature: To Low | 0 | 1 | 2 | 1 | 0
  Temperature: To w/in Range or No change | 12 | 10 | 9 | 11 | 10
  Temperature: To High | 0 | 0 | 0 | 0 | 0
  RR: To Low | 0 | 0 | 0 | 0 | 0
  RR: To w/in Range or No change | 11 | 11 | 11 | 12 | 10
  RR: To High | 1 | 0 | 0 | 0 | 0

79. Secondary Outcome: Part C: Number of Participants With Worst Case Post-Baseline Abnormal ECG Findings Following Administration of GSK3915393
Description: as for outcome 10
Time Frame: Up to 72 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK3915393 100 mcg IV | Part C: GSK3915393 100 mcg+ITZ | Part C: GSK3915393 20mg+Water | Part C: GSK3915393 20mg+GFJ | Part C: SK3915393 20 mg+ITZ
Number analyzed (Participants) | 12 | 11 | 11 | 12 | 10
Participants
  Abnormal: Not Clinically Significant | 2 | 1 | 1 | 1 | 0
  Clinically Significant | 0 | 0 | 0 | 0 | 0

80. Secondary Outcome: Part C: Number of Participants With Abnormal Physical Examination Findings Following Administration of GSK3915393
Description: as for outcome 11
Time Frame: Up to 72 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK3915393 100 mcg IV | Part C: GSK3915393 100 mcg+ITZ | Part C: GSK3915393 20mg+Water | Part C: GSK3915393 20mg+GFJ | Part C: SK3915393 20 mg+ITZ
Number analyzed (Participants) | 12 | 11 | 11 | 12 | 10
Participants | 0 | 0 | 0 | 0 | 0

81. Secondary Outcome: Part C: Fraction of Drug Escaping Hepatic Metabolism (FH) Following IV Dose of GSK3915393
Description: as for outcome 46
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1 hour 5 minutes, 1 hour 10 minutes, 1 hour 20 minutes, 1 hour 40 minutes, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 60 hours post-dose
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Ratio
Arm/Group | Part C: GSK3915393 20 mg+ Water
Number analyzed (Participants) | 11
Ratio | 0.6525 [0.435 to 0.856]

82. Secondary Outcome: Part C: FH Following IV Administration of GSK3915393+ITZ
Description: as for outcome 46
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1 hour 5 minutes, 1 hour 10 minutes, 1 hour 20 minutes, 1 hour 40 minutes, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, and 60 hours post-dose
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Ratio
Arm/Group | Part C: GSK3915393 100 mcg IV+ITZ
Number analyzed (Participants) | 11
Ratio | 0.8717 [0.780 to 0.905]

83. Secondary Outcome: Part C: Fraction of Drug Escaping Gut Metabolism (FG) Following Oral Administration of GSK3915393+Water
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393. FG was expressed as ratio and calculated as: AUC of GSK3915393+water divided by AUC of GSK3915393+GFJ.
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, and 24 hours post-dose
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Ratio
Arm/Group | Part C: GSK3915393 20 mg+ Water
Number analyzed (Participants) | 11
Ratio | NA [NA to NA] — NA indicates data is not available as estimates for FA and FG generated by analysis of the GFJ interaction study were inconsistent with pharmacokinetic data from the rest of the study and are thus not considered reliable.

84. Secondary Outcome: Part C: Fraction of Drug Absorbed (FA) Following Oral Administration of GSK3915393+Water
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3915393. FA was expressed as ratio was calculated as absolute bioavailability (F) divided by the product of fraction of drug escaping hepatic metabolism (FH) and fraction of drug escaping gut metabolism (FG).
Time Frame: Pre-dose and at 20, 40 minutes, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, and 24 hours post-dose
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Ratio
Arm/Group | Part C: GSK3915393 20 mg+ Water
Number analyzed (Participants) | 11
Ratio | NA [NA to NA] — NA indicates data is not available as estimates for FA and FG generated by analysis of the GFJ interaction study were inconsistent with pharmacokinetic data from the rest of the study and are thus not considered reliable.

ADVERSE EVENTS:
Time Frame: All-cause mortality, all non-serious and SAEs were collected up to Day 70 in Part A, up to Day 28 in Part B and up to Day 72 in Part C
Description: All-cause mortality, all non-serious AEs and SAEs were collected in Safety population comprised of all randomized participants who received at least one dose of study treatment. Placebo arms across similar dosing strategies were combined as pre-specified in reporting and analysis plan.
Arm/Group | Part A: Placebo | Part A: GSK3915393 15 mg | Part A: GSK3915393 60 mg | Part A: GSK3915393 160 mg | Part A: GSK3915393 100 mcg IV | Part B: Placebo | Part B: GSK3915393 20 mg (BID) | Part B: GSK3915393 80 mg (BID) | Part B: GSK3915393 160 mg (QD) | Part C: GSK3915393 100 mcg IV | Part C: GSK3915393 100 mcg+ITZ | Part C: GSK3915393 20 mg+ Water | Part C: GSK3915393 20 mg+ GFJ | Part C: GSK3915393 20 mg+ ITZ
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/12 | 0/10 | 0/10 | 0/9 | 0/9 | 0/12 | 0/11 | 0/11 | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/12 | 0/10 | 0/10 | 0/9 | 0/9 | 0/12 | 0/11 | 0/11 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 1/9 | 2/9 | 3/9 | 1/9 | 4/12 | 3/10 | 5/10 | 1/9 | 5/9 | 5/12 | 2/11 | 3/11 | 2/12 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=9) | Part A: GSK3915393 15 mg (N=9) | Part A: GSK3915393 60 mg (N=9) | Part A: GSK3915393 160 mg (N=9) | Part A: GSK3915393 100 mcg IV (N=12) | Part B: Placebo (N=10) | Part B: GSK3915393 20 mg (BID) (N=10) | Part B: GSK3915393 80 mg (BID) (N=9) | Part B: GSK3915393 160 mg (QD) (N=9) | Part C: GSK3915393 100 mcg IV (N=12) | Part C: GSK3915393 100 mcg+ITZ (N=11) | Part C: GSK3915393 20 mg+ Water (N=11) | Part C: GSK3915393 20 mg+ GFJ (N=12) | Part C: GSK3915393 20 mg+ ITZ (N=10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nodal rhythm (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medical device site reaction (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site bruise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Medical device site dermatitis (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Catheter site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Exposure to SARS-CoV-2 (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Cardiac telemetry traces were examined after the study had completed. For all the participants with an adverse event of ventricular tachycardia reported following repeat dosing of 160 mg QD (part B), the tracings revealed narrow QRS complex beats that "march" through the presumed wide complex beats at a fixed rate, identical to the heart rate prior to and immediately following the event. These findings support a diagnosis of artifact and are not consistent with ventricular tachycardia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial

DOCUMENTS (2):
  • Study Protocol (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT04604795/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT04604795/SAP_001.pdf